CLINICAL TRIAL: NCT05738291
Title: A Phase I Study to Assess Safety, Tolerability, Pharmacokinetics and Effect of Food on Multiple Rising Oral Doses of BI 1839100 (Single-blind, Randomised, Placebo-controlled, Parallel Group Design) and the Effect of Multiple Doses of BI 1839100 on the Single Dose Pharmacokinetics of Cytochrome P450 Substrate (Midazolam), a P Glycoprotein Substrate (Digoxin) and OATP Substrate (Rosuvastatin) Administered Orally (Open-label, Fixed-sequence) in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Well Multiple Doses of BI 1839100 Are Tolerated and How BI 1839100 Influences the Amount of Other Medicines in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1490-0002; 2022-003161-38 (EudraCT Number)
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: The multiple-rising dose (MRD) part of this trial is designed as single blinded to subject, randomised, and placebo-controlled within parallel dose groups.
  The Drug-Drug Interaction (DDI) part of this trial is designed as open-label, within-group comparison interaction trial.
Who Masked: Participant
Masking Description: MRD: single blinded to subject DDI: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- MRD part: BI 1839100 dose group 1 (Experimental): Multiple rising dose (MRD)
  Interventions: Drug: BI 1839100
- MRD part: BI 1839100 dose group 2 (Experimental): Multiple rising dose (MRD)
  Interventions: Drug: BI 1839100
- MRD part: BI 1839100 dose group 3 (Experimental): Multiple rising dose (MRD)
  Interventions: Drug: BI 1839100
- MRD part: BI 1839100 dose group 4 (Experimental): Multiple rising dose (MRD)
  Interventions: Drug: BI 1839100
- MRD part: BI 1839100 dose group 5 (Experimental): Multiple rising dose (MRD)
  Interventions: Drug: BI 1839100
- MRD part: Placebo matching BI 1839100 (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 1839100
- DDI part (Experimental): Drug-Drug Interaction (DDI)
  Interventions: Drug: BI 1839100; Drug: midazolam; Drug: digoxin; Drug: rosuvastatin

INTERVENTIONS:
Drug: BI 1839100 — BI 1839100
  Arms: DDI part; MRD part: BI 1839100 dose group 1; MRD part: BI 1839100 dose group 2; MRD part: BI 1839100 dose group 3; MRD part: BI 1839100 dose group 4; MRD part: BI 1839100 dose group 5
Drug: Placebo matching BI 1839100 — Placebo matching BI 1839100
  Arms: MRD part: Placebo matching BI 1839100
Drug: midazolam — midazolam
  Arms: DDI part
Drug: digoxin — digoxin
  Arms: DDI part
Drug: rosuvastatin — rosuvastatin
  Arms: DDI part

SUMMARY:
Effects of multiple rising doses of BI 1839100 on safety, tolerability, pharmacokinetics and the effect of high-fat meal on pharmacokinetics of BI 1839100 will be assessed as well as assessing potential drug-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 31.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm) (subjects with heart rate values between 45 and 50 bpm may only be enrolled in case they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia such as hypothyroidism or heart conduction abnormalities)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders assessed as clinically relevant by the investigator
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
MRD part: Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 26 days
  Multiple-rising dose (MRD)
DDI part: Area under the concentration-time curve of midazolam, digoxin and rosuvastatin when administered without BI 1839100 over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 20 days
  Drug-Drug Interaction (DDI)
DDI part: Maximum measured concentration of midazolam, digoxin and rosuvastatin when administered without BI 1839100 in plasma (Cmax) | up to 20 days
DDI part: Area under the concentration-time curve of midazolam, digoxin and rosuvastatin when co-administered with BI 1839100 over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 7 days
DDI part: Maximum measured concentration of midazolam, digoxin and rosuvastatin when co-administered with BI 1839100 in plasma (Cmax) | up to 7 days

SECONDARY OUTCOMES:
MRD part: Maximum measured concentration of the analyte in plasma after single dose (Cmax) | at Day 1
MRD part: Time from dosing to maximum measured concentration of the analyte in plasma (tmax) | at Day 1
MRD part: Area under the concentration-time curve of the analyte in plasma over the time interval 0 to 12 hours (AUC0-12) | at Day 1
MRD part: Area under the concentration-time curve of the analyte in plasma over the time interval 0 to 48 hours (AUC0-48) | up to 48 hours
MRD part: Area under the concentration-time curve of the analyte in plasma over a uniform 12 hours dosing interval (τ) [after Nth dose] (AUCτ( ,N)) | up to 17 days
MRD part: Maximum measured concentration of the analyte in plasma [after Nth dose] (Cmax( ,N)) | up to 17 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON-Groningen-62040, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com